CLINICAL TRIAL: NCT00898092
Title: Molecular Genetic Studies of Acute Myeloid Leukemia (AML) With Normal Cytogenetics. A CALGB Leukemia Tissue Bank Project
Brief Title: Genetics Study of Tissue Collected From Patients With Acute Myeloid Leukemia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-20502; CALGB-20502; U10CA031946 (NIH); U10CA180821 (NIH); CDR0000491133 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Leukemia
Keywords: adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7); adult acute eosinophilic leukemia; adult acute basophilic leukemia; untreated adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Basophilic, Acute | interventions — Microarray Analysis; Genetic Testing; Polymerase Chain Reaction; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Group 1: Peripheral blood and bone marrow samples are analyzed to assess gene expression using polymerase chain reaction (PCR) or reverse transcriptase-PCR assays and microarray assays. Genes to be studied include BAALC, ERB, EVI1, MLL, FLT3, NPM1, and CEBPA.
  Interventions: Genetic: microarray analysis; Genetic: molecular genetic technique; Genetic: mutation analysis; Genetic: polymerase chain reaction; Genetic: reverse transcriptase-polymerase chain reaction; Other: diagnostic laboratory biomarker analysis

INTERVENTIONS:
Genetic: microarray analysis
Genetic: molecular genetic technique
Genetic: mutation analysis
Genetic: polymerase chain reaction
Genetic: reverse transcriptase-polymerase chain reaction
Other: diagnostic laboratory biomarker analysis

SUMMARY:
RATIONALE: Collecting and storing samples of tissue and blood from patients with cancer to study in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at changes in the DNA of tissue samples that were collected from patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Validate, on the larger number of patients with karyotypically normal acute myeloid leukemia (AML) treated uniformly on CALGB-19808, preliminary results from CALGB-9621 showing that BAALC and ERG overexpression and microarray gene-expression signatures can stratify the patients prognostically.
* Establish whether microRNAs are differentially expressed in subsets of patients with AML and normal cytogenetics, and, if so, attempt to identify a signature that stratifies patients prognostically.
* Explore the relative contribution in predicting clinical outcome of patients with cytogenetically normal AML using genetic markers such as BAALC, ERG, and EVI1 overexpression, MLL partial tandem duplication, FLT3 internal tandem duplication, NPM1 and CEBPA mutations, and microarray gene expression microRNA signatures.

OUTLINE: This is a multicenter, pilot study.

Peripheral blood and bone marrow samples are analyzed to assess gene expression using polymerase chain reaction (PCR) or reverse transcriptase-PCR assays and microarray assays. Genes to be studied include BAALC, ERB, EVI1, MLL, FLT3, NPM1, and CEBPA.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia

  * Normal karyotype
* Bone marrow and/or peripheral blood samples from patients treated on CALGB-19808 and registered on CALGB-9665 required

  * No additional samples required

Ages: 15 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients enrolled on CALGB 19808 with tissue previously submitted to the CALGB Leukemia Tissue Bank
Sampling Method: Non-Probability Sample
Enrollment: 735 (Estimated)
Dates: Start 2006-05 (Actual); Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Prognostic stratification of patients through BAALC and ERG overexpression and microarray gene-expression signatures | Baseline
Differential microRNA expression | Baseline
Relative contribution of genetic markers in predicting clinical outcome | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Guido Marcucci, MD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States